CLINICAL TRIAL: NCT02544516
Title: Study on the Links Between Perception and Action in Schizophrenia, "Upside Down, Give me the Handle"
Brief Title: Upside Down, Give me the Handle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1308139; 2013-A01294-41 (Other: ANSM)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenia; motor and sensory perceptions
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): patients suffering schizophrenic disorders and who will perform cognitive tasks + PANSS+ IQ
  Interventions: Other: cognitive tasks + PANSS+ IQ
- control group (Active Comparator): healthy patients who will perform cognitive tasks
  Interventions: Other: cognitive tasks

INTERVENTIONS:
Other: cognitive tasks + PANSS+ IQ — Patients will have cognitive tasks: reaction time (Alert TEA, Zimmermann and Fimm, 2005), Edinburgh laterality questionnaire (Oldfield, 1971), IQ test (IQ: PM38, Raven, 1960), and the PANSS (Positive and Negative Syndrome Scale, Kay et al., 1987
  Arms: Patients
Other: cognitive tasks — Patients will have cognitive tasks: reaction time (Alert TEA, Zimmermann and Fimm, 2005), Edinburgh laterality questionnaire (Oldfield, 1971),
  Arms: control group

SUMMARY:
In schizophrenia, dislocation of psychic functions involving a loss of contact with reality is frequently found. A fragmentation of motor and sensory perceptions could be held responsible (Fuchs, 2005). However, automatic integration between perception and action is the necessary condition to be in "relationship with the world." Affordance is the experimental link between object perception and actions potentially associated (Gibson (1977, 1979) explored by Stimulus Response Compatibility (SRC) paradigm. The existence of visual motor neurons leads us to postulate that the affordance effect can be assisted by a visuomotor priming of a hand in a position to grasp. With Tucker & Ellis sensory motor compatibility task, we study the capacity of affordance in schizophrenia, as well as the impact of perceptual motor priming on these affordance effects.

DETAILED DESCRIPTION:
All participants will perform cognitive tasks: reaction time (Alert TEA, Zimmermann and Fimm, 2005), Edinburgh laterality questionnaire (Oldfield, 1971), IQ test (IQ: PM38, Raven, 1960), and the PANSS (Positive and Negative Syndrome Scale, Kay et al., 1987). Controls will only have the first three tasks (cognitive spots Alert and laterality). Then all will perform all tasks in successive order (task 1 and task 2). For both tasks, photographs of 20 objects of everyday life typical grip with one hand are presented in 4 orientations. The instruction is to say if the object is presented upright or inverted; The second task differs from the first only by the introduction of a prime: presenting a hand in position "catching" before the picture of an object

ELIGIBILITY:
Inclusion Criteria:

For patients:

* a DSM-IV diagnosis of schizophrenia (men or women),
* no change in antipsychotic medication and clinical status within four weeks prior to the study

Exclusion Criteria:

* IQ < 70

For patients and control group Inclusion criteria

- Age ≥ 18 years et ≤ 50 years

Exclusion Criteria:

* History of head trauma,
* neurological disease with cerebral repercussion or not stabilized serious physical illness;
* psychotropic medication,
* disorders related to the use of a psychoactive substance (abuse, dependence or withdrawal);

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
response time | day 1
  The gain provided by the compatible vs incompatible conditions (ms response time)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France